CLINICAL TRIAL: NCT04343547
Title: A Randomized, Open Label, Single/Multiple Dose, Crossover Study to Evaluate Drug-Drug Interaction of DWP16001 in Combination With DWC202001 and DWC202002 in Healthy Male Adults
Brief Title: Study to Evaluate Drug-Drug Interaction of DWP16001 in Combination With DWC202001 and DWC202002 in Healthy Male Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001104
Record Dates: First submitted 2020-04-10; First posted 2020-04-13 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — Enavogliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DWP16001
- 2 (Experimental)
  Interventions: Drug: DWC202001+DWC202002
- Experimental 3 (Experimental)
  Interventions: Drug: DWP16001+DWC202001+DWC202002

INTERVENTIONS:
Drug: DWP16001 — Tablets, Oral, once daily single dose
  Arms: 1
Drug: DWC202001+DWC202002 — Tablets, Oral, multiple doses of DWC202001 and DWC202002 in combination
  Arms: 2
Drug: DWP16001+DWC202001+DWC202002 — Tablets, Oral, DWP16001 , DWC202001 and DWC202002 in combination
  Arms: Experimental 3

SUMMARY:
The purpose of this study is to evaluate drug-drug interaction by comparing the pharmacokinetics (PK)/pharmacodynamics (PD), safety, and tolerability of single/multiple doses of DWP16001 , DWC202001 and DWC202002 alone or in combination in healthy male adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults ≥ 19 and ≤ 50 years of age at the time of the screening procedure
2. 55.0 kg ≤ body weight ≤ 90.0 kg and 18.0 ≤ body mass index (BMI) ≤ 27.0
3. Voluntarily decided to participate in the study and provided written consent prior to the screening procedure after receiving a detailed explanation on this study and fully understanding the information
4. Is eligible to participate in the study at the discretion of the investigator by a physical examination, laboratory test, and medical history questionnaire, etc.

Exclusion Criteria:

1. Presence or prior history of a clinically significant hepatic, renal, nervous, respiratory, endocrine, hematologic and oncologic, cardiovascular, urogenital, psychiatric disorder
2. Presence or prior history of a gastrointestinal disorder (e.g., gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc.), or prior history of gastrointestinal surgery (except for simple appendectomy or hernia surgery) that may affect the safety and PK/PD assessment of the study drug.
3. Hypersensitivity to, or history of clinically significant hypersensitivity to drugs including DWP16001 and other drugs of the same class (SGLT2 inhibitors), drugs including gemigliptin and other drugs of the same class, metformin and other drugs (aspirin, antibiotics, etc.)
4. Considered ineligible for the study by the investigator for reasons including laboratory test results

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cmax of DWP16001 | 0-72 hours
  Peak Plasma Concetration
AUClast of DWP16001 | 0-72 hours
  Area under the plasma concentration versus time curve
Cmax,ss of DWC202001 and DWC202002 | 0-72 hours
  Peak Plasma Concetration at steady-state
AUCτ,ss of DWC202001 and DWC202002 | 0-72 hours
  Area under the plasma concentration versus time curve at Tau, steady-state

SECONDARY OUTCOMES:
Tmax of DWP 16001, DWC202001 and DWC202002 | 0-72 hours
  Time at Cmax
T1/2 of DWP 16001, DWC202001 and DWC202002 | 0-72 hours
CL/F of DWC202001 and DWC202002 | 0-72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No